CLINICAL TRIAL: NCT01030432
Title: A Phase 2a/2b Study of BMS-650032 in Combination With Peginterferon Alfa-2a (Pegasys) and Ribavirin (Copegus) in Treatment-Naive Subjects With Genotypes 1 and 4 Chronic Hepatitis C Infection
Brief Title: Study of BMS-650032 With Peginterferon Alfa-2a Plus Ribavirin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI447-016; 2009-013652-69 (Registry Identifier: EUDRACT)
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 2a: Arm 1 (Experimental)
  Interventions: Drug: BMS-650032; Drug: Peginterferon Alfa-2a; Drug: Ribavirin
- Phase 2a: Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Peginterferon Alfa-2a; Drug: Ribavirin
- Phase 2b: Arm 1 (Experimental)
  Interventions: Drug: BMS-650032; Drug: Placebo; Drug: Peginterferon Alfa-2a; Drug: Ribavirin
- Phase 2b: Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Peginterferon Alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: BMS-650032 — Tablets, Oral, 200 mg, Twice Daily, 48 weeks
  Arms: Phase 2a: Arm 1
Drug: BMS-650032 — Tablets, Oral, 200 mg, Twice Daily, 12 or 24 weeks, depending on response
  Arms: Phase 2b: Arm 1
Drug: Placebo — Tablets, Oral, 0 mg, twice daily, 48 weeks
  Other Names: Pegasys
  Arms: Phase 2a: Arm 2
Drug: Placebo — Tablets, Oral, 0 mg, twice daily, 0 or 12 weeks (depending on response) beginning at Week 12
  Arms: Phase 2b: Arm 1
Drug: Placebo — Tablets, Oral, 0 mg, twice daily 24 weeks
  Arms: Phase 2b: Arm 2
Drug: Peginterferon Alfa-2a — Syringe, Subcutaneous injection, 180 mcg / 0.5 mL, Weekly, 48 weeks
  Other Names: Pegasys
  Arms: Phase 2a: Arm 1; Phase 2a: Arm 2; Phase 2b: Arm 2
Drug: Peginterferon Alfa-2a — Syringe, Subcutaneous injection, 180 mcg / 0.5 mL, Weekly, 24 or 48 weeks, depending on response
  Other Names: Pegasys
  Arms: Phase 2b: Arm 1
Drug: Ribavirin — Tablet, Oral, 500 or 600 mg based on weight, Twice Daily, 48 weeks
  Other Names: Copegus
  Arms: Phase 2a: Arm 1; Phase 2a: Arm 2; Phase 2b: Arm 2
Drug: Ribavirin — Tablet, Oral, 500 or 600 mg based on weight, Twice Daily, 24 or 48 weeks depending on response
  Other Names: Pegasys
  Arms: Phase 2b: Arm 1

SUMMARY:
The purpose of this study is to identify one or more doses of BMS-650032 that, when used in combination with pegylated-interferon alpha and ribavirin are safe and demonstrate sufficient activity against hepatitis C virus (Genotypes 1 and 4).

ELIGIBILITY:
Inclusion Criteria:

* Subjects chronically infected with HCV genotype 1 (Phase 2a and Phase 2b)
* Subjects chronically infected with HCV genotype 4 (Phase 2b only)
* HCV RNA viral load of ≥ 10*5* IU/mL at screening
* BMI of 18 - 35 kg/m² at screening

Exclusion Criteria:

* Cirrhosis (Phase 2a only)
* Decompensated cirrhosis (Phase 2b)
* Co-infection with HBV or HIV
* Hepatocellular carcinoma
* Prior treatment with anti-HCV drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Phase 2a and Phase 2b: Safety, as measured by the frequency of SAEs and discontinuations due to AEs | 12 weeks after first dose
Antiviral activity as determined by proportion of HCV genotype 1 subjects with extended rapid virologic response (eRVR), defined as undetectable HCV RNA | Week 4
Antiviral activity as determined by proportion of HCV genotype 1 subjects with extended rapid virologic response (eRVR), defined as undetectable HCV RNA | Week 12
Phase 2b only: Antiviral activity, as determined by the proportion of HCV genotype 1 subjects with 24-week sustained virologic response (SVR24), defined as undetectable HCV RNA | at follow-up Week 24

SECONDARY OUTCOMES:
Proportion of HCV genotype 1 subjects with rapid virologic response (RVR), defined as undetectable HCV RNA at Week 4 | Week 4
Proportion of HCV genotype 1 subjects with complete early rapid virologic response (eEVR), defined as undetectable HCV RNA at Week 12 (Stage 2 only) | at Week 12 (Stage 2 only)
Proportion of HCV genotype 1 subjects with early virologic response (EVR) defined as ≥2 log10 decrease in HCV RNA from baseline at Week 12 (Stage 1 only) | Week 12 (Stage 1 only)
Proportion of HCV genotype 1 subjects with 12-week sustained virologic response (SVR12), defined as undetectable HCV RNA at follow-up Week 12 | follow-up Week 12
Proportion of HCV genotype 1 subjects with 24-week sustained virologic response (SVR24) defined as undetectable HCV RNA at follow-up Week 24 (Stage 1 only) | follow-up Week 24 (Stage 1 only)
Resistant variants associated with virologic failure | 48 weeks after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (37):
- United States (14):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Alabama Liver & Digestive Specialists (Alds), Montgomery, Alabama
  - Florida Hospital Transplant Center, Orlando, Florida
  - Mercy Medical Center, Baltimore, Maryland
  - The Research Institute, Springfield, Massachusetts
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - James J Peters Vamc, The Bronx, New York
  - University Of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Oregon Health Science Univ, Portland, Oregon
  - Hospital Of The University Of Pennsylvania, Philadelphia, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Metropolitan Research, Fairfax, Virginia
  - Dean Clinic, Madison, Wisconsin
- Argentina (4):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Prov. Buenos Aires, Buenos Aires
  - Local Institution, Prov de Santa Fe, Santa Fe Province
- France (5):
  - Local Institution, Créteil
  - Local Institution, Marseille
  - Local Instituition, Montpellier
  - Local Institution, Paris
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (4):
  - Local Institution, Frankfurt
  - Local Institution, Heidelberg
  - Local Institution, Mainz
  - Local Institution, Würzburg
- Local Institution, Dublin, Dublin, Ireland
- Local Institution, Torino, Italy
- Spain (5):
  - Local Institution, Alicante
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Valencia
- United Kingdom (3):
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Glasgow, Lanarkshire

REFERENCES:
- [Derived] Bronowicki JP, Ratziu V, Gadano A, Thuluvath PJ, Bessone F, Martorell CT, Pol S, Terg R, Younes Z, He B, Eley T, Cohen D, Yu F, Hernandez D, McPhee F, Mendez P, Hughes E. Randomized trial of asunaprevir plus peginterferon alfa and ribavirin for previously untreated genotype 1 or 4 chronic hepatitis C. J Hepatol. 2014 Dec;61(6):1220-7. doi: 10.1016/j.jhep.2014.07.011. Epub 2014 Jul 16. PMID 25038486
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx